CLINICAL TRIAL: NCT02112955
Title: A Randomized Controlled Trial of the Effectiveness of a Nurse-led Self-efficacy Enhancing Stroke Self-management Program for Community-dwelling Stroke Survivors
Brief Title: A Self-efficacy Enhancing Stroke Self-management Program for Community-dwelling Stroke Survivors
Acronym: SESSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Suzanne Hoi-Shan Lo, PhD candidate, Queensland University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SESSMP01
Record Dates: First submitted 2014-04-09; First posted 2014-04-14 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Stroke
Keywords: Stroke; Disease management; Self efficacy; Quality of life; Community integration
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke self-management program (Experimental): The program is aimed at enhancing community-dwelling stroke survivors' post-stroke recovery.
  Interventions: Behavioral: Stroke self-management program; Behavioral: Usual care
- Usual care (Active Comparator): Usual care provided to stroke survivors discharged to their home.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Stroke self-management program — A nurse-led community-based self-efficacy enhancing stroke self-management program.
  Arms: Stroke self-management program
Behavioral: Usual care — Usual care such as hospital-based or community-based health education or services.

SUMMARY:
The aim of this study is to examine the effectiveness of a nurse-led self-efficacy enhancing stroke self-management program on recovery of community-dwelling stroke survivors.

DETAILED DESCRIPTION:
Previous systematic reviews showed that theory-based stroke self-management programs had potential benefits in improving stroke survivors' quality of life and self-efficacy. However there is a lack of evidence evaluating the effectiveness of a nurse-led theory-based stroke self-management program among community-dwelling Chinese stroke survivors.

This is a parallel group, single-blinded, randomized controlled trial to be held in a community center. All participants will be assessed at two time-points (baseline before randomization, and one month after program completion). Eligible participants will be randomly allocated to either the control group (receiving usual care) or the intervention group (receiving the self-efficacy enhancing stroke self-management program). Participants in the intervention group will receive an additional assessment on usefulness of the program immediately after program completion.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* have a clinical diagnosis of stroke
* currently live at home or will be discharged from hospital to home within one week
* have a Mini Mental State Examination score >18
* speak Cantonese
* capable of giving informed consent
* can attend sessions of the self-efficacy enhancing stroke self-management program
* can use a phone

Exclusion Criteria:

* diagnosed with transient ischemic attack, subdural or epidural hemorrhage
* have cerebrovascular events due to presence of malignancy or head trauma
* have limited comprehension and receptive aphasia
* have been diagnosed with schizophrenia, bipolar disorder, or dementia
* have received a stroke self-management program in the past 12 months as reported by the participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Self-efficacy in performing stroke self-management behaviors | One month after the program
  Stroke Self-Efficacy Questionnaire

SECONDARY OUTCOMES:
Stroke self-management behaviors | One month after the program
  Stroke Self-management Behaviors Performance Scale
Health-related quality of life | One month after the program
  Stroke Specific Quality of Life Scale
Depressive symptoms | One month after the program
  Geriatric Depression Scale
Community reintegration | One month after the program
  Reintegration to Normal Living Index
Outcome expectation | One month after the program
  Stroke Self-management Outcome Expectation Scale

OTHER OUTCOMES:
Usefulness of the program | Within one week after the completion of the program
  Extent of overall program participation, and other qualitative comments.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lo, Principal Investigator — Queensland University of Technology
Locations (3):
- Hong Kong (3):
  - Acute public hospital 1, Kowloon
  - Acute public hospital 2, New Territories
  - Acute public hospital 3, New Territories

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Lo SHS, Chang AM, Chau JPC. Stroke Self-Management Support Improves Survivors' Self-Efficacy and Outcome Expectation of Self-Management Behaviors. Stroke. 2018 Mar;49(3):758-760. doi: 10.1161/STROKEAHA.117.019437. Epub 2018 Feb 2. PMID 29438073
- [Derived] Lo SH, Chang AM, Chau JP. Study protocol: a randomised controlled trial of a nurse-led community-based self-management programme for improving recovery among community-residing stroke survivors. BMC Health Serv Res. 2016 Aug 15;16(a):387. doi: 10.1186/s12913-016-1642-9. PMID 27528049